CLINICAL TRIAL: NCT04696094
Title: The Role of m6A RNA Modification in Moyamoya Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY 2020-118-03
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Moyamoya Disease
Keywords: m6A
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Health volunteers' inclusion criteria:
  Age between 4-60; Male or female;
  Exclusion criteria:
  Exclude the volunteers with history of cerebrovascular disease.
- Moyamoya disease patients: Moyamoya disease patients' inclusion Criteria:
  1.written informed consent had been obtained; 2. more than 4 years old and less than 60 years old; 3. cerebral digital subtraction contrast angiography (DSA) revealed severe stenosis or occlusion of the distal internal carotid or proximal middle and anterior cerebral arteries with prominent lenticulostriate 'moyamoya collaterals'; 4. received surgical revascularization;
  Exclusion Criteria:
  1. There are other vascular diseases, including systemic vasculitis, neurofibroma, meningitis, sickle cell disease, down's syndrome, and previous basilar radiotherapy; 2. Patients with cardiogenic embolism, including a history of atrial fibrillation, valvular disease or cardiac valve replacement; 3. Physical or subjective failure to cooperate with the examination or serious comorbid diseases.

SUMMARY:
The purpose of this study is to detect the change of m6A RNA modification from peripheral blood of patients with moyamoya disease, and to assess the relationship between clinical characteristics.

DETAILED DESCRIPTION:
Moyamoya disease (MMD) is a rare cerebrovascular disorder characterized by occlusion of bilateral internal carotid and intracerebral arteries with the compensatory growth of fragile small vessels. The etiology of disease is still unclear. The pathology is associated with blood vessels, characterizing the molecular changes of blood in patients with MMD may yield insights into the disease. N6-methyladenosine (m6A) is identified to be the most common and abundant RNA molecular modification in eukaryotes, and involves in a variety of metabolic processes of RNA, such as RNA transcription, shearing, nuclear transport, and translation ability. The propose of this study is to investigate the change of m6A RNA modification in patients blood with moyamoya disease and its influence on clinical indicators, aiming to provide potential pathogenesis of moyamoya disease.

ELIGIBILITY:
Health volunteers' inclusion criteria:

Age between 4-60; Male or female;

Exclusion criteria:

Exclude the volunteers with history of cerebrovascular disease.

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Moyamoya disease patients
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
m6A RNA modification in peripheral blood | 2021.1.1-2021.12.31
  m6A RNA modification in peripheral blood

SECONDARY OUTCOMES:
Suzuki grade | 30days
  Stage 1 stenosis of the carotid artery at its suprasellar portion, usually bilateral; Stage 2 moyamoya vessels begin to develop at the base of the brain; Stage 3 moyamoya vessels become more prominent as major trunks in the anterior circulation become severely stenotic or occluded; Stage 4 posterior cerebral arteries are occluded, moyamoya vessels begin to diminish and collateral pathways from extracranial circulation develop; Stage 5, moyamoya vessels are diminishing and extracranial circulation progresses; Stage 6, moyamoya vessels and the major cerebral arteries completely disappear, the cerebral hemispheres receive blood through the abnormal extracranial-intracranial anastomosis.
  Higher scores mean a worse outcome.
Modified Rankin Scale score | 6months
  0 No symptoms at all; 1 No significant disability despite symptoms, able to carry out all usual duties and activities; 2 Slight disability, unable to carry out all previous activities, but able to look after own affairs without assistance; 3 Moderate disability, requiring some help, but able to walk without assistance; 4 Moderately severe disability, unable to walk without assistance and unable to attend to own bodily needs without assistance; 5 Severe disability, bedridden, incontinent and requiring constant nursing care and attention.
  Higher scores mean a worse outcome.
New clinical vascular events | 6 months
  New clinical vascular events (ischemic stroke/ hemorrhagic stroke/ TIA)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No